CLINICAL TRIAL: NCT02399917
Title: An Open-Label Phase II Study of Lirilumab (BMS-986015) in Combination With 5-Azacytidine (Vidaza) for the Treatment of Patients With Refractory/Relapsed Acute Myeloid Leukemia
Brief Title: Lirilumab and Azacitidine in Treating Patients With Refractory or Relapsed Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated early due to response rates not meeting the anticipated minimum of 30%.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0862; NCI-2015-00678 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0862 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Acute Biphenotypic Leukemia; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Acute | interventions — Azacitidine; lirilumab

STUDY DESIGN:
Intervention Model Description: Phase IB, lead-in/II to determine MTD
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1b Lead-in Cohort 1 (Experimental): Patients receive azacitidine SC or IV over 1 hour as determined by the treating physician on days 1-7 and lirilumab IV over 60 minutes on day 8. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  5-Azacitidine 75mg/m^2 Lirilumab 1.0 mg/kg
  Interventions: Drug: Azacitidine; Biological: Lirilumab
- Phase 1b Lead-in Cohort 2 (Experimental): Patients receive azacitidine SC or IV over 1 hour as determined by the treating physician on days 1-7 and lirilumab IV over 60 minutes on day 8. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  5-Azacitidine 75mg/m^2 Lirilumab 3.0 mg/kg
  Interventions: Drug: Azacitidine; Biological: Lirilumab
- Phase 2 (Experimental): Patients receive azacitidine SC or IV over 1 hour as determined by the treating physician on days 1-7 and lirilumab IV over 60 minutes on day 8. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  5-Azacitidine 75mg/m^2 Lirilumab 3.0 mg/kg
  Interventions: Drug: Azacitidine; Biological: Lirilumab

INTERVENTIONS:
Drug: Azacitidine — Given SC or IV
  Other Names: 5 AZA; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Biological: Lirilumab — Given IV
  Other Names: BMS-986015; IPH2102

SUMMARY:
This phase II trial studies the side effects lirilumab and azacitidine and to see how well they work in treating patients with acute myeloid leukemia that has not responded to treatment or has returned after a period of improvement. Monoclonal antibodies, such as lirilumab, may interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving lirilumab with azacitidine may be an effective treatment for relapsed or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of lirilumab in combination with 5-azacytidine (azacitidine) in patients with refractory/relapsed acute myeloid leukemia (AML). (Part A, Lead-In Phase) II. To determine the overall response rate (ORR) of lirilumab in combination with 5-azacytidine in patients with refractory/relapsed AML. (Part B, Phase II)

SECONDARY OBJECTIVES:

I. To determine the duration of response, disease-free survival (DFS), and overall survival (OS) of patients with refractory/relapsed AML treated with this combination.

II. To determine the safety of lirilumab in combination with 5-azacytidine in patients with refractory/relapsed AML.

OUTLINE:

Patients receive azacitidine subcutaneously (SC) or intravenously (IV) over 1 hour as determined by the treating physician on days 1-7 and lirilumab IV over 60 minutes on day 8. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and up to 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML or biphenotypic or bilineage leukemia who have failed at least one prior therapy; patients with AML should have failed prior therapy or have relapsed after prior therapy
* Patients should not be eligible or able to receive approved therapy of confirmed clinical benefit in this patient population
* Patients with myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia (CMML) who received therapy for the MDS or CMML and progress to AML are eligible at the time of diagnosis of AML regardless any prior therapy for AML; the World Health Organization (WHO) classification will be used for AML
* Prior therapy with hydroxyurea, chemotherapy, biological or targeted therapy (e.g. FLT3 inhibitors, other kinase inhibitors), or hematopoietic growth factors is allowed
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin =< 2 times upper limit of normal (x ULN) (=< 3 x ULN if considered to be due to leukemic involvement or Gilbert's syndrome)
* Aspartate aminotransferase or alanine aminotransferase =< 2.5 x ULN (=< 5.0 x ULN if considered to be due to leukemic involvement)
* Serum creatinine =< 2 x ULN or glomerular filtration rate (GFR) >= 50
* Patients must provide written informed consent
* In the absence of rapidly progressing disease, the interval from prior treatment to time of initiation of 5-azacytidine and lirilumab will be at least 2 weeks OR at least 5 half-lives for cytotoxic/noncytotoxic agents; use of one dose of cytarabine (up to 2 g/m^2) is allowed prior to the start of study therapy or hydroxyurea for patients with rapidly proliferative disease is allowed before the start of study therapy and while the patient is on active study treatment, as needed, for clinical benefit and after discussion with the principal investigator (PI); concurrent therapy for central nervous system (CNS) prophylaxis or continuation of therapy for controlled CNS disease is permitted
* Females must be surgically or biologically sterile or postmenopausal (amenorrheic for at least 12 months) or if of childbearing potential, must have a negative serum or urine pregnancy test within 72 hours before the start of the treatment
* Women of childbearing potential must agree to use an adequate method of contraception during the study and until 30 days after the last treatment; males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 30 days after the last treatment; women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago; in the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential

Exclusion Criteria:

* Patients with known allergy or hypersensitivity to lirilumab, 5-azacytidine, or any of their components; patients who have previously been treated with lirilumab in combination with 5-azacytidine will be excluded
* Patients with a known history of severe interstitial lung disease or severe pneumonitis or active pneumonitis that is uncontrolled in the opinion of the treating physician
* Patients with a known history of any of the following autoimmune diseases are excluded: (a) patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) (b) patients with a history of rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis])
* Patients with organ allografts (such as renal transplant) are excluded
* Patients with allogeneic stem cell transplantation within the last 6 months or patients with active graft-versus-host disease (GVHD) will be excluded
* Ongoing immunosuppressive therapy, including cyclosporine and tacrolimus; patients who are on high dose steroid; Note: Subjects may be using systemic corticosteroids (daily doses =< 10 mg of prednisone or equivalent) or topical or inhaled corticosteroids
* Patients with symptomatic CNS leukemia or patients with poorly controlled CNS leukemia
* Active and uncontrolled disease/(active uncontrolled infection, uncontrolled hypertension despite adequate medical therapy, active and uncontrolled congestive heart failure New York Heart Association [NYHA] class III/IV, clinically significant and uncontrolled arrhythmia) as judged by the treating physician
* Patients with active and uncontrolled human immunodeficiency virus (HIV) infection will be excluded; however, patients with well controlled HIV infection will be considered
* Patients known to be positive for hepatitis B by surface antigen expression; known to have active hepatitis C infection (positive by polymerase chain reaction or on antiviral therapy for hepatitis C within the last 6 months)
* Any other medical, psychological, or social condition that may interfere with study participation or compliance, or compromise patient safety in the opinion of the investigator
* Patients unwilling or unable to comply with the protocol
* Pregnant or breastfeeding
* Acute promyelocytic leukemia (APL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naval Daver, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 2015 - June 2017
Groups:
- Phase 1b Lead-in Cohort 1: Patients receive azacitidine SC or IV over 1 hour as determined by the treating physician on days 1-7 and lirilumab IV over 60 minutes on day 8. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  5-Azacitidine 75mg/m^2 Lirilumab 1.0 mg/kg
  Azacitidine: Given SC or IV
  Lirilumab: Given IV
- Phase 1b Lead-in Cohort 2; Phase 2: Patients receive azacitidine SC or IV over 1 hour as determined by the treating physician on days 1-7 and lirilumab IV over 60 minutes on day 8. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  5-Azacitidine 75mg/m^2 Lirilumab 3.0 mg/kg
  Azacitidine: Given SC or IV
  Lirilumab: Given IV
Period: Overall Study
Arm/Group | Phase 1b Lead-in Cohort 1 | Phase 1b Lead-in Cohort 2 | Phase 2
Started | 6 | 6 | 24
Completed | 6 | 6 | 24
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b Lead-in Cohort 1 | Phase 1b Lead-in Cohort 2 | Phase 2 | Total
Number analyzed (Participants) | 6 | 6 | 24 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 13 | 20
  >=65 years | 2 | 3 | 11 | 16
Age, Continuous [Median (Full Range); unit: years] | 59.5 [48 to 84] | 68.5 [32 to 89] | 65 [30 to 76] | 64 [30 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 14 | 18
  Male | 5 | 3 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 4 | 5
  White | 5 | 6 | 19 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 24 | 36

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Iirilumab in Combination With 5-azacitidine
Description: To identify the dose at which <2/6 participants experience Dose Limiting Toxicities (DLT). The dose level at which 0-1/6 participants experience a DLT in the first 28 days of treatment will be the maximum tolerated dose (MTD) and would be used to treat an additional 34 participants in the phase II potion of the study. (Part A, Lead-In Phase)
Time Frame: Up to 28 days
Measure: Number; unit: mg/kg
Groups:
- All Phase 1 Participants: Patients receive azacitidine SC or IV over 1 hour as determined by the treating physician on days 1-7 and lirilumab IV over 60 minutes on day 8. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  5-Azacitidine 75mg/m^2 Lirilumab 1.0 mg/kg
  Azacitidine: Given SC or IV
  Lirilumab: Given IV
Arm/Group | All Phase 1 Participants
Number analyzed (Participants) | 12
mg/kg | 3.0

2. Primary Outcome: Participants With an Objective Response
Description: Objective Response Rate (ORR) will be monitored using the Bayesian approach of Thall, Simon, Estey and the extension by Thall and Sung. Overall response rate (ORR), defined as complete remission (CR) + CR with incomplete platelet recovery (CRp) + CR with incomplete count recovery (CRi) + partial response (PR) + marrow clearance of blasts + hematological improvement within 3 months of treatment initiation among adult patients with refractory/relapsed Acute Myelogenous Leukemia (AML) (Phase II)
Time Frame: Up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Lead-in Cohort 1 | Phase 1b Lead-in Cohort 2 | Phase 2
Number analyzed (Participants) | 6 | 6 | 24
Participants | 2 | 1 | 2

3. Secondary Outcome: Duration of Response
Description: The date of Objective Response to the date of loss of response or last follow-up.
Time Frame: Up to 2.5 years
Population: The outcome for the secondary response, duration of response was only done on the Phase II portion of this study.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 1b Lead-in Cohort 1 | Phase 1b Lead-in Cohort 2 | Phase 2
Number analyzed (Participants) | 0 | 0 | 24
Months |  |  | 7.7 [2.0 to 17.0]

4. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is defined: Time of presentation to date of death or censored at last follow-up date.
Time Frame: Up to 2 years
Population: The outcome for the secondary response, overall response was only done on the Phase II portion of this study.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 1b Lead-in Cohort 1 | Phase 1b Lead-in Cohort 2 | Phase 2
Number analyzed (Participants) | 0 | 0 | 24
Months |  |  | 3.5 [0.4 to 22.2]

5. Secondary Outcome: Disease Free Survival
Description: Disease Free Survival (DFS) is defined: Time from date of treatment start until the date of first objective documentation of disease-relapse
Time Frame: Up to 2.5 years
Population: The outcome for the secondary response, disease free survival was only done on the Phase II portion of this study.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 1b Lead-in Cohort 1 | Phase 1b Lead-in Cohort 2 | Phase 2
Number analyzed (Participants) | 0 | 0 | 24
Months |  |  | 7.7 [2.0 to 17.0]

ADVERSE EVENTS:
Time Frame: Up to two and a half years.
Arm/Group | Phase 1b Lead-in Cohort 1 | Phase 1b Lead-in Cohort 2 | Phase 2
All-Cause Mortality (participants affected / at risk) | 4/6 | 2/6 | 9/24
Serious Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 20/24
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 22/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b Lead-in Cohort 1 (N=6) | Phase 1b Lead-in Cohort 2 (N=6) | Phase 2 (N=24)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Blood and Lymphatic system disorders (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenic Fever (Infections and infestations) | 2 (3) | 2 (3) | 9 (19)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Disorders Other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileal Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 2 (2) | 4 (8)
Joint Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 4 (5) | 0 (0) | 10 (16)
Mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Multi-Organ Failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Respiratory other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Scrotal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 3 (4)
Skin Infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Spinal Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Surgical/medical procedures other (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b Lead-in Cohort 1 (N=6) | Phase 1b Lead-in Cohort 2 (N=6) | Phase 2 (N=24)
Abdominal Distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0)
Elevated Alanine Aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Aspartate Aminotransferase Increased (Investigations) | 2 (2) | 3 (3) | 4 (4)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3)
Constipation (Gastrointestinal disorders) | 1 (2) | 1 (1) | 10 (12)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 8 (8)
Edema (General disorders) | 1 (1) | 1 (1) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 5 (5)
Fever (General disorders) | 3 (3) | 0 (0) | 8 (9)
Headache (General disorders) | 2 (2) | 0 (0) | 3 (3)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4)
Hyperbilirubinemia (Investigations) | 1 (1) | 1 (1) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 3 (3)
Hypomagnesmia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 8 (8)
Infection (Infections and infestations) | 2 (2) | 0 (0) | 7 (8)
Infusion Reaction (General disorders) | 1 (1) | 1 (1) | 7 (11)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 4 (4)
Mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4)
Neutropenic Fever (Infections and infestations) | 3 (3) | 0 (0) | 6 (6)
Pain (General disorders) | 1 (1) | 2 (4) | 10 (16)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 0 (0) | 5 (5)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 7 (7)
Pneumonia (Infections and infestations) | 3 (5) | 2 (2) | 4 (4)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 6 (7)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 7 (9)
Weight Loss (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT02399917/Prot_SAP_000.pdf